CLINICAL TRIAL: NCT05430685
Title: The Impact of Ashwagandha on Stress, Sleep and Food Cravings in College Students: A Mixed Method Double-blinded Randomized Control Trial
Brief Title: The Impact of Ashwagandha on Perceived Stress, Sleep and Food Cravings in College Students
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Colorado, Colorado Springs (Other)
Responsible Party: Principal Investigator, Margaret Harris, Associate Professor, University of Colorado, Colorado Springs
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 19-132
Record Dates: First submitted 2022-05-27; First posted 2022-06-24 (Actual); Last update posted 2022-06-24 (Actual); Status verified 2022-06

CONDITIONS: Stress; Sleep; Craving; Well Being
Keywords: Ashwagandha
MeSH Terms: interventions — Ashwagandha; Glycerol

STUDY DESIGN:
Intervention Model Description: Two groups: one intervention, one placebo
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The company (Gaia Herbs) prepared the intervention and placebo and had knowledge with Intervention A and B. Neither the investigators, coordinators, subjects or data analyst had knowledge of the group designation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ashwagandha (Experimental): Generic name: ashwagandha root extract Dose form: Chloroform capsule Dose: 1 capsule 350 mg ashwagandha root extract Frequency: 2 times per day (one capsule in the morning, one capsule in the evening). Total: 700 mg ashwagandha root extract per day Duration: 30 days
  Interventions: Dietary Supplement: Ashwagandha
- Placebo (Placebo Comparator): Generic name: placebo Dose form: Glycerin equivalent weight to ashwagandha Dose: 1 capsule Frequency: one capsule, 2 times per day (one capsule in morning and one in evening) Duration: 30 dys
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Ashwagandha — Intervention and placebo group each received a bottle of 60 capsules. Subjects were instructed to take one capsule in the morning and 1 capsule in the evening. Intervention group was getting 350 mg ashwagandha root extract per capsule (or 700 mg per day). Each intervention capsule delivered 2.5 mg withanolides with equivalence of 2,700 mg dry herb.
  Other Names: Gaia Herbs; Withania somnifera
  Arms: Ashwagandha
Other: Placebo — The Placebo group received the same type of bottle with similar looking capsules. Each person in the placebo group was instructed to take 1 capsule twice a day (2 capsules total). Capsules were filled with glycerin to the same weight as ashwagandha. Capsules were indistinguishable from each other.
  Other Names: glycerin
  Arms: Placebo

SUMMARY:
The purpose of this study was to compare the impact of 700 mg daily ashwagandha (Withania Somnifera) in healthy college students on sleep, stress and food cravings to healthy college students taking placebo.

DETAILED DESCRIPTION:
College aged students tend to report significant daily stress but there is no research on herbal interventions to ameliorate this condition in this population.

This study is a mixed methods, randomized, double blinded, placebo controlled 30 day trial targeting a college aged population. Participants are randomly allocated to either an intervention group (ashwagandha) or a placebo group. Each participant is given a bottle of capsules (capsules look identical but are filled either with a full spectrum dried extract ashwagandha herb or a placebo filled with glycerin). Directions included consuming 1 capsule in the morning and one capsule in the evening. Questionnaires were collected prior to the study and at the end of the study, including an assessment of daily affect. A subset of each group volunteered to attend an intervention specific focus group at 30 days completion of the study.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older
* Enrolled at the university

Exclusion Criteria:

* sensitivity to nightshade vegetables;
* peptic ulcer;
* pregnant or expected to become pregnant in the near future;
* breastfeeding;
* had recent or planned surgery;
* hypotensive;
* diagnosed with diabetes;
* and/or taking any of the following classes of medications: benzodiazepines, central nervous system depressants, diabetes medication, thyroid medication, immune suppressors, cardiovascular medication.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — People of any gender identity were eligible
Enrollment: 60 (Actual)
Dates: Start 2019-05-29 (Actual); Primary Completion 2020-04-10 (Actual); Study Completion 2020-04-10 (Actual)

PRIMARY OUTCOMES:
Impact of ashwagandha on Sleep | Change of restorative sleep quality at 30 days
  Restorative Sleep Questionnaire is a 9-item validated scale assessing feelings and experiences about the participant's sleep and their perception of daytime consequences associated with their sleep patterns. Scores range from 0-100 where higher scores indicate better quality sleep.
Impact of ashwagandha on Perceived Stress | Change of perceived stress at 30 days
  Stress was assessed using the Perceived Stress Scale a 10-item validated questionnaire measuring the degree to which situations in participant's life were viewed as stressful. Questions addressed anxious thoughts, locus of control, and coping mechanisms. Scores range from 0-40 (higher scores indicate higher stress levels).
Impact of ashwagandha on Food Cravings | Change of food cravings at 30 days
  Eating behavior was assessed using the Food Cravings Questionnaire, a 15-item validated instrument assessing food behavior and appetite using Likert-scales related to intentions for eating, perceived control, hunger cues, emotional states, and guilt associated with cravings. Scores range between 15 and 90 (higher scores indicate more frequent and intense food cravings).

SECONDARY OUTCOMES:
Qualitative analysis of ashwagandha on college students across sleep, stress and food cravings. | At 30 days
  A virtual focus group conducted with each intervention group separately and was recorded via a video conferencing platform. Transcript was downloaded and investigators read for thematic analysis.
Daily check in qualitative analysis | Up to 30 days
  Participants checked in via Microsoft Teams private chat with a daily question "How are you doing today?" Transcripts were downloaded and analyzed using a qualitative analysis software for coding and thematic analysis

CONTACTS AND LOCATIONS:
Overall Officials: Margaret Harris, PhD, Principal Investigator — University of Colorado, Colorado Springs
Locations (1):
- University of Colorado Colorado Springs, Colorado Springs, Colorado, United States

REFERENCES:
- [Derived] O'Connor J, Lindsay K, Baker C, Kirby J, Hutchins A, Harris M. The Impact of Ashwagandha on Stress, Sleep Quality, and Food Cravings in College Students: Quantitative Analysis of a Double-Blind Randomized Control Trial. J Med Food. 2022 Dec;25(12):1086-1094. doi: 10.1089/jmf.2022.0040. Epub 2022 Aug 18. PMID 35984871
- [Derived] Baker C, Kirby JB, O'Connor J, Lindsay KG, Hutchins A, Harris M. The Perceived Impact of Ashwagandha on Stress, Sleep Quality, Energy, and Mental Clarity for College Students: Qualitative Analysis of a Double-Blind Randomized Control Trial. J Med Food. 2022 Dec;25(12):1095-1101. doi: 10.1089/jmf.2022.0042. Epub 2022 Aug 18. PMID 35984870